CLINICAL TRIAL: NCT06604416
Title: Acute Effect of Forward and Backward Walking Exercise on Physical and Cognitive Functions
Brief Title: Forward and Backward Walking Exercise on Physical and Cognitive Functions
Status: Completed | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Hilal Denizoğlu Külli, Assoc. Prof, Atlas University
Other Study IDs: edaserenkarakaya
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers
Keywords: backward walking; aerobic exercise; cognitive functions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Backward walking exercise group: Healthy subjects aged 18-25 years were included in the study. Cognitive and physical function assessments were performed face-to-face by a physiotherapist before and after backward walking exercise. In addition, assessments during the exercise were performed by the same physiotherapist. Assessments were made immediately before and immediately after the walking exercise. All assessments were supervised by the physiotherapist.
  Interventions: Other: Backward walking
- Forward walking exercise group: Healthy subjects aged 18-25 years were included in the study. Cognitive and physical function assessments were performed face-to-face by a physiotherapist before and after forward walking exercise. In addition, assessments during the exercise were performed by the same physiotherapist. Assessments were made immediately before and immediately after the walking exercise. All assessments were supervised by the physiotherapist.
  Interventions: Other: Forward walking
- Control group: Participants did not perform any walking exercise. Cognitive and physical function assessments were performed before and after the assessment tests, with 30 minutes of rest in between.

INTERVENTIONS:
Other: Forward walking — The exercises consisted of a 5-minute warm-up on a treadmill followed by a 25-minute period of moderate forward walking.
  Groups: Forward walking exercise group
Other: Backward walking — The exercises consisted of a 5-minute warm-up on a treadmill followed by a 25-minute period of moderate backward walking.
  Groups: Backward walking exercise group

SUMMARY:
To investigate the acute effects of forward and backward walking exercise on physical functions such as static and dynamic balance and cognitive functions such as attention, concentration, memory, processing speed, visual structuring skills, calculation and orientation.

DETAILED DESCRIPTION:
This study is planned to investigate the acute effects of forward and backward walking on physical functions such as static and dynamic balance and cognitive functions such as attention, concentration, memory, processing speed, visual structuring skills, calculation and orientation. 50 healthy individuals were randomly divided into three groups for the study. The groups were divided into Backward Walking Exercise Group (GYE) (n=17), Forward Walking Exercise Group (FWE) (n=16) and Control Group (CG)(n=17). Before treatment for all three groups; sociodemographic and clinical data with the sociodemographic information form, physical activity levels with the International Physical Activity Survey Short Form, pain severity with the Visual Analog Scale (VAS), fatigue levels with the Borg Scale, the person's selective attention capacity and skills, processing speed and general executive processing abilities. Stroop Test with TBAG Form to evaluate executive functions such as working memory, complex attention, planning and set shifting, with Trail Making Test, evaluation of dynamic balance, neuromuscular control and movement asymmetries with Y-Balance Test, static balance, postural stability evaluation on One Leg It was evaluated with the Standing Test. The GYE group completed a 25-minute backward walking exercise session, the FWE group completed a 25-minute forward walking exercise session, and the control group completed a 30-minute sitting rest between evaluation tests. After the exercises, there were significant differences in parameters such as attention, processing speed, concentration and maintenance of attention, working memory, planning, static and dynamic balance, and in the comparison between groups, significant differences were found in static balance and postural control (p<0.05). It was observed that individuals in the backward walking group showed better improvements in some parameters after walking. However, these results need to be supported by future studies.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-25,
* To be able to communicate verbally and in written Turkish,
* Not complaining of pain in any part of the body during physical activity,
* Performing a normal walking pattern without compensatory movements.

Exclusion Criteria:

* Participants participating in a routine exercise program
* History of upper or lower extremity pathology or injury in the last 6 months
* Diagnosed neurological disease
* Diagnosed cognitive impairment
* Having a diagnosed orthopedic disease
* Using a walking aid
* Inadequate cardiovascular fitness
* Dyspnea on exertion
* Contraindication to walking
* Receiving medical treatment that causes imbalance.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy university students aged 18-25 years were included in the study, excluding physically active individuals according to the International Physical Activity Scale Short Form.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Stroop Test TBAG Form | immediately pre and immediately post-exercise
  Stroop Test TBAG Form was used to assess executive functions such as attention, memory, concentration, visual structuring skills, computational working memory, planning, visual scanning ability.
Trail Making Test | immediately pre and immediately post-exercise
  The Trail Making Test was used to assess executive functions such as working memory, complex attention, planning and set switching, visual-spatial processing and motor abilities. The Trail Making Test consists of two parts, A and B.
Y-Balance Test | immediately pre and immediately post-exercise
  Y-Balance Test was used to evaluate dynamic balance, neuromuscular control and movement asymmetries.
One Leg Standing Test | immediately pre and immediately post-exercise
  One-leg Standing Test was used to assess static balance.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) Short Form | pre-assessments
  The IPAQ Short Form was used to determine the physical activity levels of the participants.
The Visual Analog Scale (VAS) | immediately pre and immediately post-exercise
  This scale scores from 0 to 10. Higher scores indicate worse pain.
Borg Fatigue Scale | immediately pre-exercises, during exercise and immediately post-exercise
  It was used to determine the level of fatigue perceived by individuals before, during and after completing walking exercises.
Oxygen Saturation | immediately pre-exercises, during exercise and immediately post-exercise
  In the study, saturation values were measured by pulse oximetry before, during and after exercise by the same physiotherapist.
Blood Pressure Assessment | immediately pre and immediately post-exercise
  Blood pressure assessment was performed with a syphinguometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Kagıthane, Turkey (Türkiye)